CLINICAL TRIAL: NCT04252495
Title: An Open-label Phase 1 Study to Investigate the Effect of Moderate Hepatic Impairment Due to Liver Cirrhosis on the Pharmacokinetics of a Single Dose of 25 mg Aprocitentan
Brief Title: The Effect of Hepatic Impairment on Aprocitentan Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-080-109; 2019-003580-21 (EudraCT Number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Hepatic Impairment; Healthy Subjects
Keywords: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — aprocitentan

STUDY DESIGN:
Intervention Model Description: Healthy subjects will be matched to subjects with moderate hepatic impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with moderate hepatic impairment (Group 1) (Experimental)
  Interventions: Drug: Aprocitentan
- Healthy subjects (Group 2) (Experimental)
  Interventions: Drug: Aprocitentan

INTERVENTIONS:
Drug: Aprocitentan — A single oral dose of 25 mg.
  Other Names: ACT-132577

SUMMARY:
This is a prospective, open-label, single-dose, Phase 1 study, to assess the effect of moderate hepatic impairment due to liver cirrhosis on the pharmacokinetics of aprocitentan (ACT-132577).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Women of childbearing potential (WoCBP) must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1 and must agree to use highly effective methods of contraception from screening up to 30 days after study treatment.
* A Women of non-childbearing potential (WoNCBP) must meet one of the following criteria:

  * Previous bilateral salpingectomy, salpingo-oophorectomy or hysterectomy.
  * Premature ovarian failure confirmed by a specialist gynecologist.
  * Post-menopausal, defined as 12 consecutive months with amenorrhea prior to screening without alternative medical cause and confirmed with a follicle stimulating hormone test.
* Body mass index of 18.0 to 35.0 kg/m2 (inclusive) at screening.
* Normal renal function confirmed by a creatinine clearance at screening according to Cockcroft and Gault adjusted to age.
* Additional principal inclusion criteria for subjects with moderate hepatic impairment (Group 1)

  * Moderate hepatic function impairment due to liver cirrhosis defined as a score of 7-9 (inclusive) according to the Child-Pugh classification.
  * Systolic blood pressure 95 to 160 mmHg, diastolic blood pressure 60 to 95 mmHg, and pulse rate 50 to 100 bpm (inclusive), measured on the same arm, after 5 minutes in the supine position at screening and on Day 1 pre-dose.
  * International normalized ratio equal or less than 2.5 at screening.
  * Stable concomitant medications for at least 3 weeks prior to screening and up to Day 1 and expected to be stable during the conduct of the study.
* Additional principal inclusion criteria for healthy subjects (Group 2)

  * Healthy on the basis of medical history, physical examination, cardiovascular assessments, and clinical laboratory tests.

Exclusion Criteria:

* Pregnant or lactating women.
* Previous exposure to aprocitentan and/or macitentan.
* Known hypersensitivity to any excipients of the drug formulation.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Any signs or symptoms of active, ongoing infection judged to be clinically relevant by the investigator (special attention should be given to COVID-19, e.g., fever, dry cough, dyspnea, sore throat, or fatigue).
* Subjects must adhere to the clinical site's house rules, which include, amongst others, polymerase chain reaction testing for SARS-CoV-2 at screening and admission.
* Legal incapacity or limited legal capacity at screening.
* Additional exclusion criteria for subjects with moderate hepatic impairment (Group 1)

  * History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion (ADME) of the study treatment except for those related to liver cirrhosis (appendectomy and herniotomy allowed, cholecystectomy not allowed).
  * Hepatic cancer, primary biliary cirrhosis, or any form of cholestatic disease.
  * Clinical evidence or suspected acute liver failure as judged by the investigator.
  * Encephalopathy grade greater than 2.
  * Severe ascites and/or pleural effusion.
  * Clinically relevant findings in clinical laboratory tests (hematology, coagulation, clinical chemistry, and urinalysis) at screening & on Day -1, except for those related to liver cirrhosis.
* Additional exclusion criteria for healthy subjects (Group 2)

  * Clinically relevant findings on the physical examination at screening.
  * History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion (ADME) of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed).
  * Clinically relevant findings in clinical laboratory tests (hematology, coagulation, clinical chemistry, and urinalysis) at screening & on Day -1.
  * Clinically relevant abnormalities on a 12-lead ECG, recorded after 5 min in the supine position at screening & on Day 1 pre-dose.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of aprocitentan | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 14.
Area under the plasma concentration-time curves (AUC0-t) of aprocitentan | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 14.
Area under the plasma concentration-time curve to infinity (AUC0 to inf) of aprocitentan | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 14.

SECONDARY OUTCOMES:
Treatment-emergent Adverse Events | From study treatment administration on Day 1 up to last assessment on End of Study (Day 15)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (2):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany
- Biokinetica S.A., Józefów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fontes MSC, Dingemanse J, Halabi A, Tomaszewska-Kiecana M, Sidharta PN. Single-dose pharmacokinetics, safety, and tolerability of the dual endothelin receptor antagonist aprocitentan in subjects with moderate hepatic impairment. Sci Rep. 2022 Nov 9;12(1):19067. doi: 10.1038/s41598-022-22470-z. PMID 36352054